CLINICAL TRIAL: NCT01061801
Title: Emotional Expression and Cancer Caregivers
Brief Title: Spouses/Partners Expressing Their Thoughts After Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Shelby Langer (Principal Investigator), Fred Hutchinson Cancer Research Center and the University of Washington
Allocation: Randomized | Masking: None | Purpose: Basic Science
Other Study IDs: 2076.00
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Cancer; Hematopoietic Stem Cell Transplantation
Keywords: caregivers; cancer; emotion; protective buffering
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Emotional expression, patient present (Experimental): Caregivers are asked to talk about their deepest thoughts and feelings regarding the patient's transplant and their role as caregiver, in the presence of the patient (one session).
  Interventions: Behavioral: Emotional expression
- Emotional expression, patient absent (Experimental): Caregivers are asked to talk about their deepest thoughts and feelings regarding the patient's transplant and their role as caregiver, in the absence of the patient (3 sessions).
  Interventions: Behavioral: Emotional expression
- Comparison (Active Comparator): Caregivers are asked to talk about their plans for the upcoming week (time management, sessions 1 and 3) and positive aspects of their life (session 2).
  Interventions: Behavioral: Emotional expression

INTERVENTIONS:
Behavioral: Emotional expression — Caregivers are given the opportunity to express their thoughts and feelings regarding the patient's transplant and their role as caregiver
  Other Names: Emotional disclosure

SUMMARY:
This study seeks to test a brief psychological intervention for spousal caregivers of cancer patients (specifically, hematopoietic stem cell transplant patients), persons known to experience emotional distress.

DETAILED DESCRIPTION:
This project focuses on spousal caregivers (CGs) of hematopoietic stem cell transplant survivors - persons known to report elevated levels of distress as compared to both norms and their patient counterparts. Specific Aims are to: (1) Determine, via experimental manipulation, whether or not CGs of hematopoietic stem cell transplant patients engage in protective buffering, a coping mechanism whereby partners shield patients from illness-related concerns or worries, (2) Examine synchrony or lack thereof, desynchrony, among subjective, expressive and biologic indicators of emotion among spousal CGs, and (3) Test the feasibility and implementation of an emotional expression (EE) exercise designed to enhance psychological and immune functioning among spousal CGs.

ELIGIBILITY:
Inclusion Criteria:

* patients and partners at least 21 years of age
* patients and partners English speaking
* patients about to receive a hematopoietic stem cell transplant
* patients married or in a committed, cohabiting, heterosexual or homosexual relationship
* caregivers in a married or committed, cohabiting, heterosexual or homosexual relationship with the patient
* caregivers present at the transplant site and planning to remain so for at least one month

Exclusion Criteria:

* patient major psychiatric disorder
* caregiver presence or history of a neurologic disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Self-reported mental and physical health as measured by the Short Form-36 Health Survey | baseline, 1-month follow-up, and 4-month follow-up
Marital satisfaction as measured by the Dyadic Adjustment Scale | pre-transplant, baseline, 1-month follow-up, and 4-month follow-up
Self- and partner-reported protective buffering as measured by the Protective Buffering Scale | pre-transplant, baseline, 1-month follow-up, and 4-month follow-up

SECONDARY OUTCOMES:
Emotional experience as assessed by the Positive and Negative Affect Schedule | During intervention/ disclosure sessions
Galvanic skin response (physiological indicator of emotion) | During intervention/ disclosure sessions
Emotional expression (facial expression and words uttered) | During intervention/ disclosure sessions

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Langer, PhD, Principal Investigator — FHCRC/UW Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Langer SL, Brown JD, Syrjala KL. Intrapersonal and interpersonal consequences of protective buffering among cancer patients and caregivers. Cancer. 2009 Sep 15;115(18 Suppl):4311-25. doi: 10.1002/cncr.24586. PMID 19731352